CLINICAL TRIAL: NCT05072314
Title: Long-term Outcomes of Lidocaine Infusions for Post-Operative Pain (LOLIPOP) Trial
Acronym: LOLIPOP
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Monash University (Other)
Collaborators: Royal Perth Hospital (Other)
Responsible Party: Principal Investigator, Prof Tomas Corcoran, Chief Principal Investigator, Monash University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HREC/74777/Alfred-2021
Record Dates: First submitted 2021-10-03; First posted 2021-10-08 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer; Breast Cancer Female; Breast Conserving Surgery; Mastectomy
Keywords: Anaesthesia; Local Anaesthesia; Chronic Post Surgical Pain
MeSH Terms: conditions — Breast Neoplasms; Pain, Postoperative | interventions — Lidocaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All trial participants, research coordinators, members of the anaesthesia and surgical teams, pharmacists, theatre and ward staff and all individuals performing patient follow up will be blinded to the patient's treatment allocation. All of the trial committees associated with the study will be blinded, with the exception of the Data Safety and Monitoring Committee (DSMC), who will receive unblinded (open) reports from the independent statistician. Unblinding of the patient's treatment allocation will be possible in exceptional circumstances, and a process will be in place to facilitate unblinding requests.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lidocaine (Active Comparator): 2% Lidocaine infusion intra-operative and 10% Lidocaine infusion post-operative.
  Interventions: Drug: lidocaine 2% and 10%
- Placebo (Placebo Comparator): 0.9% Saline infusion intra-operative and 0.9% Saline infusion post-operative.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: lidocaine 2% and 10% — Lidocaine infusion:
  1. Commencing with an intravenous bolus after induction of anaesthesia, 0.125 ml/kg of lean body weight (LBW) of 2% lidocaine (2.5 mg/kg).*
  2. Followed by a 2% lidocaine intravenous infusion for the duration of surgery, 0.1665 ml/kg/h of LBW (3.33 mg/kg/hr).*
  3. A post-operative subcutaneous 0.0222 ml/kg/hr of LBW 10% lidocaine infusion for up to 24 hours thereafter (2.22 mg/kg/hr). Dosage will be capped at a maximum lean body weight of 68kg.
     * *Day-case surgery receives intraoperative bolus and intraoperative infusion only
  Other Names: Xylocaine (lidocaine) 2% and Xylocard (lidocaine) 10%
  Arms: Lidocaine
Drug: Placebo — Placebo infusion:
  1. Commencing with an intravenous bolus after induction of anaesthesia, 0.125 ml/kg of lean body weight (LBW) of 0.9% Saline solution.*
  2. Followed by a 0.9% Saline solution intravenous infusion for the duration of surgery, 0.1665 ml/kg/h of LBW (3.33 mg/kg/hr).*
  3. A post-operative subcutaneous 0.0222 ml/kg/hr of LBW 0.9% Saline solution infusion for up to 24 hours thereafter (2.22 mg/kg/hr). Dosage will be capped at a maximum lean body weight of 68kg.
     * *Day-case surgery receives intraoperative bolus and intraoperative infusion only
  Other Names: 0.9% Saline solution
  Arms: Placebo

SUMMARY:
The LOLIPOP Trial is a large (n=4,300 patients) pragmatic, international, multicentre, prospective, randomised, double blind, placebo-controlled, parallel assessment, safety and effectiveness superiority study.

DETAILED DESCRIPTION:
The Trial's purpose is to evaluate the effectiveness of lidocaine infusions commenced during surgery and extending up to 24 hours postoperatively, on the incidence of moderate or severe chronic post-surgical pain (CPSP) detected one year following surgery in female patients undergoing elective breast cancer surgery. The trial has 90% power to detect a clinically meaningful (25%) reduction in the incidence of the primary outcome. Secondary outcomes include safety events, analgesic efficacy (pain scores and opioid consumption), neuropathic characteristics of CPSP, and psychological and quality of life outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Consenting adult female patients (≥18 years) undergoing mastectomy (unilateral or bilateral) or breast conserving surgery (unilateral or bilateral) for the primary excision of confirmed or suspected primary breast cancer under general anaesthesia (including those with simultaneous insertion of tissue expanders or implants)*. * this specifically excludes patients undergoing surgery for locoregional recurrence
* American Society of Anaesthesiologist (ASA) physical scale 1-3

Exclusion Criteria:

* Mastectomy or breast conserving surgery with add on procedures e.g laparoscopic salpingectomy
* Where surgery is being performed for locoregional recurrence of breast cancer
* Pre-existing pain at site of surgery, axilla, ipsilateral side of chest wall or the ipsilateral upper arm (at diagnosis prior to any tumor locating procedures)
* Re-excision procedures where the margins at the index surgery have been deemed insufficient
* When immediate autologous reconstruction surgery is planned
* Where delayed autologous reconstruction surgery on the operative breast within one year is planned
* Planned use of regional analgesia infusions
* Impaired cognition
* Pregnant or lactating females
* Transgender patients
* Known metastatic disease
* History of anaphylaxis, sensitivity or known contraindication to lidocaine (or other amide local anaesthetic agents e.g. other amide local anaesthetic agents: ropivacaine, bupivacaine, mepivacaine, prilocaine, etidocaine), including patients with porphyria or methaemoglobinaemia
* History of epilepsy
* Baseline heart rate < 50 bpm or systolic blood pressure < 100mmHg.
* Acute coronary event in the last three months
* Cardiac conduction abnormalities, including; Atrial fibrillation, Heart block (all degrees), Bundle Branch Block or Fascicular block, Prolonged QT interval, Wolf Parkinson White syndrome, channelopathy such as Brugada syndrome. A preoperative Electrocardiogram (ECG) is not mandatory, unless clinically indicated
* Abnormal serum potassium concentration (based upon site laboratory reference ranges)
* Active liver disease e.g. viral hepatitis, alcoholic liver disease, non-alcoholic fatty liver disease, haemochromatosis, other rarer causes)
* Medications within the last 7 days which are known / suspected to slow lidocaine metabolism (amiodarone, beta blockers, cimetidine, fluoroquinolones, fluvoxamine, imidazoles, macrolides, verapamil, HIV drugs)
* Cardiac Failure (any documented heart failure at peroperative assessment or GP records)
* Severe Renal Failure (Creatinine Clearance of less than 30ml/min or dialysis dependent)
* Co-administration of lidocaine within 24 hours prior to surgery for other reasons (e.g. lidocaine patches

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 4300 (Estimated)
Dates: Start 2022-07-27 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
The incidence of moderate or severe CPSP at 1 year after surgery, as reported by the patient at the follow-up review. | 1 year post-surgery
  Numerical rating scale ≥4 out of 10 for worst pain in the last week - The pain must have been present for at least 3 months prior to the one year assessment (or longer).

SECONDARY OUTCOMES:
The incidence of severe CPSP at 1 year after surgery | 1 year post surgery
  NRS for worst pain the in the last week of ≥7)
Severity of pain at the site of surgery | 1 year post surgery
  Assessed using "average" and "worst" NRS pain score in the last week, obtained from the adapted modified Brief Pain Inventory-Short Form (mBPI-SF)
Incidence of neuropathic symptoms | 1 year post surgery
  Incidence examined as a binary outcome using the Short Form of Douleur Neuropathique 4 Questions (S-DN4)
Physical functioning | 1 year post surgery
  Using interference component of mBPI-SF
Changes in quality of life metrics EuroQol 5 Dimension 5 Level (EQ-5D-5L) at 1 year after surgery compared to baseline | 1 year post surgery
  Changes in the quality of life
Changes in psychological wellbeing Kessler Psychological Distress Scale (K-10) at 1 year after surgery compared to baseline. | 1 year post surgery
  Changes in psychological wellbeing
The incidence of mild or greater pain at the site of surgery at 1 year after surgery | 1 year post surgery
  NRS for worst pain the in the last week of ≥1
The incidence of discomfort or altered sensation at the site of surgery (not reported as pain) | 1 year post surgery
  Patients asked if they have any altered sensation at the site of surgery
Severity of acute postoperative pain at rest | 24 hours postoperatively
  Maximum pain score, Numerical rating scale (NRS) 0-10
Severity of Acute postoperative pain on movement | 24 hours postoperatively
  Maximum pain score, Numerical rating scale (NRS) 0-10
Postoperative opioid consumption | on Day 1
  Morphine Equivalent Opioid Consumption (MEQ)
Postoperative opioid consumption | 3 months (last 24-hours)
  Morphine Equivalent Opioid Consumption (MEQ)
Postoperative opioid consumption | 1 year post surgery (last 24 hours)
  Morphine Equivalent Opioid Consumption (MEQ)
The incidence of mortality at 1 year | 1 year post surgery
  Mortality at 1 year
UK NHS costs of care over 1 year following surgery | 1 year post surgery
  UK/NHS sites only
Productivity costs over 1 year following surgery | 1 year post surgery
  UK/NHS sites only
Quality-adjusted life years (QALYs) over 1 year following surgery | 1 year post surgery
  UK/NHS sites only
Cost-effectiveness of perioperative lidocaine infusions compared to usual care, from a primary UK NHS perspective and broader perspective including productivity, at 1 year. | 1 year post surgery
  UK/NHS sites only

OTHER OUTCOMES:
Incidence of treated bradycardia intraoperatively | 24 hours postoperatively
  Drug related safety Endpoints
Incidence of treated hypotension intraoperatively | 24 hours postoperatively
  Drug related safety Endpoints
Incidence of treated bradycardia in Post Anaesthesia Care Unit (PACU) | 24 hours postoperatively
  Drug related safety Endpoints
Incidence of treated hypotension in Post Anaesthesia Care Unit (PACU) | 24 hours postoperatively
  Drug related safety Endpoints
Incidence of intraoperative infusion stopping events | 24 hours postoperatively
  Drug related safety Endpoints
Incidence of Post Anaesthesia Care Unit (PACU) infusion stopping events | 24 hours postoperatively
  Drug related safety Endpoints, (x2 symptoms, x1 sign, x1 complication)
Incidence of postoperative infusion stopping events on the ward | 24 hours postoperatively
  Drug related safety Endpoints, (x2 symptoms, x1 sign, x1 complication)
Incidence of suspected lidocaine toxicity events | 24 hours postoperatively
  Drug related safety Endpoints
Incidence of suspected SEVERE lidocaine toxicity events | 24 hours postoperatively
  Drug related safety Endpoints, (generalised seizure, sudden unexplained LOC, life-threatening arrhythmia, or asystole, cardiac or circulatory arrest)
Incidence of Medical Emergency Team (MET) activation | 24 hours postoperatively
  Drug related safety Endpoints
Incidence of unplanned Intensive Care Unit (ICU), High Dependency Unit (HDU) or Critical Care Unit (CCU) admission | 24 hours postoperatively
  Drug related safety Endpoints
Incidence of study drug unblinding events | 24 hours postoperatively
  Drug related safety Endpoints
Incidence of subcutaneous catheter site events | Day 30
  Drug related safety Endpoints

CONTACTS AND LOCATIONS:
Overall Officials: Tomas Corcoran, Principal Investigator — Royal Perth Hospital
Locations (45):
- Australia (25):
  - Blacktown Mount Druitt Hospital, Mount Druitt, New South Wales
  - Royal North Shore Hospital, Sydney, New South Wales
  - Westmead Hospital, Sydney, New South Wales
  - St George Hospital, Sydney, New South Wales
  - Royal Brisbane and Women's Hospital, Brisbane, Queensland
  - Queen Elizabeth II Jubilee Hospital, Coopers Plains, Queensland
  - Mackay Base Hospital, Mackay, Queensland
  - Rockhampton Hospital, Rockhampton, Queensland
  - Gold Coast Hospital and Health Service- Gold Coast University Hospital, Southport, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Flinders Medical Centre, Bedford Park, South Australia
  - Royal Hobart Hospital, Hobart, Tasmania
  - Anaesthetic Group Ballarat, Ballarat, Victoria
  - Ballarat Health Services (Grampians Health), Ballarat, Victoria
  - Barwon Health - University Hospital Geelong, Geelong, Victoria
  - The Alfred, Melbourne, Victoria
  - Royal Melbourne Hospital, Melbourne, Victoria
  - St Vincent's Hospital Melbourne, Melbourne, Victoria
  - Northern Hospital, Melbourne, Victoria
  - Monash Health - Moorabbin Hospital, Melbourne, Victoria
  - Maroondah Hospital - Eastern Health, Ringwood East, Victoria
  - Goulburn Valley Health, Shepparton, Victoria
  - Latrobe Regional Hospital, Traralgon, Victoria
  - Royal Perth Hospital, Perth, Western Australia
  - St John of God Subiaco, Perth, Western Australia
- Hong Kong (3):
  - North District Hospital, Shatin, Sha Tin
  - Pamela Youde Nethersole Eastern Hospital, Chai Wan
  - Ruttonjee Hospital, Wan Chai
- New Zealand (3):
  - Auckland City Hospital, Auckland, Auckland
  - Middlemore Hospital, Auckland, Middlemore
  - Waikato Hospital, Hamilton, Waikato Region
- United Kingdom (14):
  - University Hospital Wishaw, Wishaw, Scotland
  - Belfast City Hospital, Belfast
  - Southmead Hospital, North Bristol Trust, Bristol
  - Darlington Memorial Hospital, Darlington
  - Russells Hall Hospital, Dudley
  - Royal Liverpool and Broadgreen Hospitals, Liverpool
  - Whittington Hospital, London
  - Royal Marsden Hospital, London
  - Newcastle upon Tyne Hospitals, Newcastle upon Tyne
  - Norfolk and Norwich University Hospital, Norwich
  - Rotherham NHS Foundation Trust, Rotherham
  - University Hospital Southampton, Southampton
  - St Helen's Hospital, St Helens
  - Torbay Hospital, Torquay

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Toner AJ, Bailey MA, Schug SA, Corcoran TB. A pilot multicentre randomised controlled trial of lidocaine infusion in women undergoing breast cancer surgery. Anaesthesia. 2021 Oct;76(10):1326-1341. doi: 10.1111/anae.15440. Epub 2021 Mar 2. PMID 33651896
- [Background] Toner AJ, Bailey MA, Schug SA, Phillips M, Ungerer JP, Somogyi AA, Corcoran TB. Serum lidocaine (lignocaine) concentrations during prolonged perioperative infusion in patients undergoing breast cancer surgery: A secondary analysis of a randomised controlled trial. Anaesth Intensive Care. 2023 Nov;51(6):422-431. doi: 10.1177/0310057X231194833. Epub 2023 Oct 6. PMID 37802488